CLINICAL TRIAL: NCT05788991
Title: Comparative Study of the Efficacy and Safety of Vaginally Applied Dequalinium Chloride (10 mg) and Orally Applied Metronidazole (2 x 500 mg) in the Treatment of Bacterial Vaginosis
Brief Title: Comparison of Dequalinium Chloride (Fluomizin) vs Oral Metronidazole for the Treatment of Bacterial Vaginosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Medinova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MNFM380119; 2020-002489-15 (EudraCT Number)
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-06

CONDITIONS: Bacterial Vaginosis; Vaginal Infection; Vaginal Diseases
Keywords: bacterial vaginosis; dequalinium chloride; metronidazole; vaginal infection treatment; comparative study; non inferiority
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginitis; Vaginal Diseases | interventions — Dequalinium; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dequalinium chloride (Experimental): Dequalinium chloride 10 mg vaginal tablets
  Interventions: Drug: Dequalinium Chloride
- Metronidazole (Active Comparator): Metronidazole 500 mg oral tablets
  Interventions: Drug: Metronidazole Oral

INTERVENTIONS:
Drug: Dequalinium Chloride — Fluomizin vaginal tablets (10 mg dequalinium chloride) used once a day for 6 days
  Other Names: Fluomizin
  Arms: Dequalinium chloride
Drug: Metronidazole Oral — Metronidazole oral tablets (500 mg) taken twice a day for 7 days
  Arms: Metronidazole

SUMMARY:
The goal of this clinical trial is to show the efficacy and safety of dequalinium chloride in the treatment of bacterial vaginosis compared to metronidazole.

DETAILED DESCRIPTION:
Eligible patients who signed informed consent were randomized to receive treatment with either dequalinium chloride (+ oral placebo) or metronidazole (+ vaginal placebo) for up to 7 days. Primary objective was clinical cure rate at one week after start of treatment. Control visits to assess outcomes were done after end of treatment and after one month.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal woman ≥18 years
2. Diagnosis of bacterial vaginosis (all 4 Amsel criteria positive, i.e. 1) greyish white thin discharge, 2) postassium hydroxide (KOH) test or 'fishy' smell, 3) microscopic presence of > 20% clue cells, 4) vaginal pH > 4.5)
3. Signed Written Informed Consent to participate in this study

Exclusion Criteria:

1. Pregnancy and/or lactation based on urine Pregnancy test (women with childbearing potential should use any contraception excluding vaginal methods like vaginal ring, etc.)
2. Uterine bleeding (including menstruation) or vaginal bleeding of unknown origin
3. Ulcerations/erosions of vaginal mucosa or cervix uteri
4. Patients with clinical symptoms and findings of Candida vulvovaginitis and/or Aerobic vaginitis
5. Clinically manifest or suspicion of sexually transmitted infections (Neisseria gonorrhoeae, Chlamydia trachomatis, or Trichomonas vaginalis) based on signs, symptoms, and anamnesis
6. Use of any antimicrobial treatment (local or systemic) 14 days before entry the study
7. Use of any vaginal medication or vaginal douching 7 days before entry the study
8. Unwillingness to refrain from alcohol consumption during treatment, and 48 hours after treatment
9. Severe systemic diseases (HIV, cancer, tuberculosis, autoimmune diseases, diabetes mellitus, severe psychiatric conditions, etc.), including diseases treated with immunosuppressive therapies, systemic corticosteroids, or warfarin
10. Known or suspected hypersensitivity to one of the study medications, inclusive of their excipients
11. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant (including inability to fill-in electronic patient diary)
12. Participation of patient in another investigational drug study concomitantly or within 30 days prior to entry in the study
13. Patient is relative of, or staff directly reporting to, the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Grob, PhD, Study Director — Medinova AG
Locations (14):
- Czechia (4):
  - Centrum ambulantní gynekologie a primární péče, s.r.o., Brno
  - G-CENTRUM Olomouc s.r.o., Olomouc
  - Gynekologicko-porodnická ambulance, Ústí nad Labem
  - GYNEKO spol. s r.o, Vsetín
- Poland (5):
  - Salve Medica Sp. z o. o. S. K., Lodz
  - NZOZ All-Med Centrum Medyczne, Lodz
  - 1 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ, Lublin
  - KO-MED CENTRA KLINICZNE Sp. z o.o. Ośrodek, Lublin
  - Prywatny Gabinet Ginekologiczno-Położniczy, Żurawica
- Slovakia (5):
  - GPN, s.r.o., Bratislava
  - RADMA GYN s.r.o., Bratislava
  - GYNEDUR s.r.o, Dubnica nad Váhom
  - MCM GYNPED s.r.o., Dubnica nad Váhom
  - GYNECARE s.r.o., Púchov

REFERENCES:
- [Result] Raba G, Durkech A, Malik T, Bassfeld D, Grob P, Hurtado-Chong A; Fluomizin Study Group. Efficacy of Dequalinium Chloride vs Metronidazole for the Treatment of Bacterial Vaginosis: A Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e248661. doi: 10.1001/jamanetworkopen.2024.8661. PMID 38696172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: July 2021 to August 2022
Period: Overall Study
Arm/Group | Dequalinium Chloride | Metronidazole
Started (Randomized) | 73 | 78
Completed (Completed 1 month follow up) | 70 | 72
Not Completed | 3 | 6
Not completed — Not treated with study medication | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Population: Randomized= 151 patients but 4 did not receive study medication because of consent withdrawal (1 for dequalinium chloride, 3 for metronidazole) Received intervention= 147 (72 dequalinium chloride, 75 metronidazole) but 4 were missing the primary outcome assessment (3 for dequalinium chloride and 1 for metronidazole) Patients with data for primary endpoint analysis= 147 (69 dequalinium chloride, 74 metronidazole)
Groups:
- Total: Total of all reporting groups
Arm/Group | Dequalinium Chloride | Metronidazole | Total
Number analyzed (Participants) | 72 | 75 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (9.2) | 37.5 (8.9) | 36.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 75 | 147
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 72 | 75 | 147
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Nugent Score [Count of Participants; unit: Participants] — Nugent score uses a 0 to 10 scale: 0 - 3 = normal flora, 4 - 6 = intermediate flora, 7 - 10 = bacterial vaginosis
  Participants
    Normal | 18 | 23 | 41
    Intermediate | 15 | 10 | 25
    Bacterial vaginosis | 39 | 41 | 80
    Missing score | 0 | 1 | 1
Vaginal infections in the last 12 months [Median (Inter-Quartile Range); unit: events] | 1.0 [0 to 3.0] | 0 [0 to 3.0] | 1 [0 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate
Description: Resolution of the abnormal vaginal discharge, negative whiff test, and less than 20% clue cells
Time Frame: One week after randomization (C1)
Population: Patients who were randomized, treated, and with primary outcome data available
Measure: Count of Participants; unit: Participants
Arm/Group | Dequalinium Chloride | Metronidazole
Number analyzed (Participants) | 69 | 74
Participants | 64 | 69
Statistical Analysis 1: Comparison: Dequalinium Chloride vs Metronidazole; The outcome measure of the primary objective was a noninferiority margin of 15 percentage points in the absolute difference in clinical cure rates between dequalinium chloride and metronidazole 7 to 11 days after start of treatment; Test type: Non-Inferiority — Difference of proportions between groups (with 95% CI) and a non inferiority margin of 15 percentage points, assuming a 1-sided α = .025 and 80% power; p < .025, Farrington-Manning test — 1 sided alpha; Farrington-Manning test = -0.5, 95% CI 1-sided [lower limit -10.8]

2. Secondary Outcome: Clinical Cure Rate
Description: Resolution of the abnormal vaginal discharge, negative whiff test, and less than 20% clue cells
Time Frame: One month after randomization (C2)
Measure: Number; unit: participants
Arm/Group | Dequalinium Chloride | Metronidazole
Number analyzed (Participants) | 69 | 71
participants | 55 | 62

3. Secondary Outcome: Bacteriological Cure Rate
Description: Nugent score ≤3
  Nugent score uses a 0 - 10 scale (higher score mean a worse outcome): 0 - 3 = normal flora, 4 - 6 = intermediate flora, 7 - 10 = bacterial vaginosis
Time Frame: One week & one month
Population: Some patients were missing the Nugent score
Measure: Count of Participants; unit: Participants
Arm/Group | Dequalinium Chloride | Metronidazole
Number analyzed (Participants) | 69 | 74
Participants
  Visit 1 (1 week) | 35 | 51
  Visit 2 (1 month): number analyzed (Participants) | 69 | 71
  Visit 2 (1 month) | 28 | 38

4. Secondary Outcome: Therapeutic Cure
Description: Combination of clinical and bacteriological cure
Time Frame: One week & one month
Population: Some patients had a missing Nugent score
Measure: Count of Participants; unit: Participants
Arm/Group | Dequalinium Chloride | Metronidazole
Number analyzed (Participants) | 69 | 74
Participants
  Visit 1 (1 week) | 34 | 48
  Visit 2 (1 month): number analyzed (Participants) | 69 | 71
  Visit 2 (1 month) | 26 | 33

5. Secondary Outcome: Subjective Assessment of Efficacy
Description: Efficacy was assessed by patients and investigators as 'very good', 'good', 'moderate' or 'poor'.
Time Frame: One week
Population: Many missing values
Measure: Count of Participants; unit: Participants
Arm/Group | Dequalinium Chloride | Metronidazole
Number analyzed (Participants) | 69 | 74
Participants
  Investigator: Very Good | 46 | 49
  Investigator: Good | 18 | 20
  Investigator: Moderate | 4 | 4
  Investigator: Poor | 1 | 1
  Patient: number analyzed (Participants) | 50 | 54
  Patient: Very Good | 19 | 22
  Patient: Good | 26 | 24
  Patient: Moderate | 4 | 8
  Patient: Poor | 1 | 0

6. Secondary Outcome: Subjective Assessment of Tolerability
Description: Tolerability was assessed by patients as 'very good', 'good', 'moderate' or 'poor'.
Time Frame: One week
Population: Many missing values
Measure: Count of Participants; unit: Participants
Arm/Group | Dequalinium Chloride | Metronidazole
Number analyzed (Participants) | 50 | 54
Participants
  Very good | 30 | 21
  Good | 17 | 26
  Moderate | 3 | 4
  Poor | 0 | 3

7. Post Hoc Outcome: Patients Cured Based on Standard Amsel Criteria
Description: Amsel criteria = presence of abnormal vaginal discharge, whiff test (fishy odor), clue cells, and pH >4.5 Bacterial vaginosis = 3 or more Amsel criteria present Cure = absence of 2 or more Amsel criteria
Time Frame: 1 week and 1 month
Population: Missing some outcome measures
Measure: Count of Participants; unit: Participants
Arm/Group | Dequalinium Chloride | Metronidazole
Number analyzed (Participants) | 69 | 74
Participants
  One week | 68 | 73
  One month: number analyzed (Participants) | 69 | 71
  One month | 61 | 67

ADVERSE EVENTS:
Time Frame: 1 month
Description: Safety population included patients who received treatment with study medication (dequalinium chloride or metronidazole). Treatment-emergent adverse events, defined as adverse events occurring within 24 days of randomization.
Arm/Group | Dequalinium Chloride | Metronidazole
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/75
Other Adverse Events (participants affected / at risk) | 4/72 | 10/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dequalinium Chloride (N=72) | Metronidazole (N=75)
Candidiasis (Reproductive system and breast disorders) | 2 (2) | 4 (4)
vaginal infection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal burnining sensation (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pruritus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal swelling (General disorders) | 2 (2) | 0 (0)
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT05788991/Prot_SAP_000.pdf